CLINICAL TRIAL: NCT03381820
Title: Instrumental Folk Music Listening Reduced Home Blood Pressure in Stage-2 Hypertensive Patients; a Randomized Controlled Trial
Brief Title: Effectiveness of Thai Northeastern Folk Musical Therapy for Blood Pressure Control in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Principal investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE581320
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Musical Therapy as a Complementary Treatment of Hypertension
Keywords: music therapy; hypertension; Asian; stage-2 hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomised control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music listening (Experimental): Participants who were randomized into intervention group were assigned to listen to the music everyday (day 1st to day 30th), at anytime of day that was suitable with their lifestyles but not at the time of BP measurement. During day 31st -120th, participants did not listen to the music. Other treatment was the same as the control arm.
  Interventions: Other: instrumental folk music
- control (No Intervention): control arm received conventional hypertension treatment.

INTERVENTIONS:
Other: instrumental folk music — The music was composed and edited by a professor of Folk Musical Department, Faculty of Arts, Khon Kaen University. There were total of 6 songs, 32-minute length. The music was slow-instrumental, 60-80 beats per minute and ranged between 40-60 decibel levels.
  Arms: music listening

SUMMARY:
A randomized controlled trial was conducted in a tertiary care hospital, Khon Kaen province, Thailand. Sixty participants were randomized to music listening group and control group. The music listening group was assigned to listen to 30-minute instrumental folk music everyday for one month. Home BP and office BP were monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old
* Diagnosed stage-2 hypertension (HT) (defined by office systolic blood pressure >= 140mm Hg and/or diastolic blood pressure >= 90 mm Hg at first hospital visit)

Exclusion Criteria:

* Pregnant women, white-coat HT, secondary HT and hearing loss or blind.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline of home systolic and diastolic blood pressure at day 30th | Day 0th (baseline) to day 30th.
  Home blood pressure of participant was monitored and recorded.

SECONDARY OUTCOMES:
Change from baseline of office systolic and diastolic blood pressure at day 120th | Day 0th and day 120th
  Office blood pressure was measured at day 0th (baseline) and at day 120th (3-month follow up).

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Medicine, Khon Kaen University, Khon Kaen, Muang, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data is available when contact and request to the correspondence author or principal investigator.

REFERENCES:
- [Derived] Im-Oun S, Kotruchin P, Thinsug P, Mitsungnern T, Techa-Atik P, Pongchaiyakul C. Effect of Thai instrumental folk music on blood pressure: A randomized controlled trial in stage-2 hypertensive patients. Complement Ther Med. 2018 Aug;39:43-48. doi: 10.1016/j.ctim.2018.05.014. Epub 2018 May 26. PMID 30012391